CLINICAL TRIAL: NCT04673838
Title: The Effect of Lower Limb Sensory Training on Functional Capacity in Hemiparetic Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Gulsum Tikac, Principal Investigator, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hemiparetic Sensory Training
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2021-03

CONDITIONS: Hemiparesis/Hemiplegia (One Sided Weakness/Paralysis)
MeSH Terms: conditions — Paresis; Hemiplegia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lower Extremity Sensory Training + Bobath Therapy (Experimental): Intervention Group will have Lower extremity sensory training and Bobath Therapy.
  Interventions: Other: neurodevelopmental therapy; Other: Lower extremity sensory training
- Bobath Therapy (Active Comparator): Control Group will have only Bobath Therapy. Bobath approach will be applied for 4 weeks, 3 days a week and 12 sessions in total.
  Interventions: Other: neurodevelopmental therapy

INTERVENTIONS:
Other: neurodevelopmental therapy — Considering the individual needs and wishes of the patient, an exercise program will be created for each patient in accordance with their functional levels and supporting active participation of the person. The treatment program tailored to the patient; It will include weight transfer to the affected side in different positions, functional reaching out activities, stepping forward and walking activities.
  Other Names: Bobath Therapy
Other: Lower extremity sensory training — Lower extremity sensory training will only be applied to the Intervention Group for 4 weeks, 3 days a week and 12 sessions in total. In the lower extremity, 3 sets of soft tissue needing, stroking and fascia stretching will be applied on 5 areas as Quadriceps, Hamstring, Gastrosoleus Group, Peroneal muscles, ankle and foot. In addition, sensory stimulation will be applied in the same five regions of the lower extremity with 3 repetitions and 3 sets with a knurled ball, brush and sponge. Lower extremity mobilizations of PANat Therapy approach will be used with traction and gliding applications in all joints in the ankle and foot. Finally, intrinsic muscle stimulation will be performed for 3 minutes with a bottle and towel under the sole of the foot.
  Arms: Lower Extremity Sensory Training + Bobath Therapy

SUMMARY:
The purpose of our study is to assess the effect of lower limb sensory training on proprioception, balance, gait and motor functions in Hemiparetic Individuals.

DETAILED DESCRIPTION:
After being informed about the study, all patients giving written informed consent will be determined eligibility for study entry. Patients who meet the eligibility requirements will be randomized in a single-blind manner (investigor about assessments). A group will have Bobath Therapy and the other group Bobath and Sensory Training.

ELIGIBILITY:
Inclusion Criteria: for Intervention and Control Group:

* Between the ages of 20-65 and discharged from the hospital,
* Having been diagnosed with hemiparesis at least 4 weeks ago,
* First time and one-sided hemiparesis,
* Modified Rankin Score ≤3,
* Hodkinson Mental Test ≥ 6,
* Individuals who agree to having treatment will be included in the study.

Exclusion Criteria:for Intervention and Control Group:

* Having vision and hearing problems,
* Having other neurological, psychiatric and / or orthopedic problems other than hemiparesis,
* Medically unstable,
* Have other diagnosed diseases that will affect lower extremity sensation,
* Individuals with open wounds, circulatory problems, skin lesions in the area to be treated will be excluded from the study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-12-20 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Functional Level | 4 weeks
  Motricity Index (MI) will be used to determine motor function levels. Since the lower extremity functions after hemiparesis are evaluated in the study, the lower extremity score of the Motricity Index will be calculated. In the lower extremity, hip flexion muscle strength, knee extension muscle strength, and ankle dorsi flexion muscle strength will be evaluated in the sitting position. Each muscle is evaluated over 33. The highest score obtained from the test is 100 and shows the best functionality.
Foot Sole Sense | 4 weeks
  he evaluation will be done with Semmes Weinstein Monofilaments (SWM) in the supine position. Monofilaments will be held perpendicular to the surface, and they will be contacted for 1.5-2 seconds by pressing until there is a slight bend in the monofilament. Individuals will be informed to say "yes" when they feel the contact, and the responses obtained from the patient will be recorded. The application will be evaluated in seven regions on the sole of the foot: the big toe, the little toe, the first metatarsal, the fifth metatarsal, the lateral border of the foot, the medial border of the foot, and the medial border of the heel. Thicknesses in the test kit range have from 1.65 to 6.55. The 6.65 is the loss of protective sensation and is the worst result.
Lower Extremity Position Test | 4 weeks
  It was developed for the evaluation of proprioseption after stroke. Two 12 cm and 22 cm lines are drawn in the middle of the A4 paper. The patient is seated on a flat chair and the toes are adjusted to match the tip of the paper. The eyes of the patient are closed, the tips of the toes are brought over the line twice passively, and in the next evaluation, the patient is informed about "stop" and the difference is recorded in cm. The smaller is the difference, the better is proprioseption.
Kinesthesia Sense | 4 weeks
  Measurement will be done with electrogoniometer in the sitting position. 60 degrees hip flexion, 60 degrees knee flexion and 10 degrees ankle plantar flexion angles will be performed on the healthy leg in 5 repetitions, then three measurements will be taken from the hemiparetic leg.
Balance Assessment | 4 weeks
  The device consists of two parts, an electronic inclination sensor and a moving platform. There is a red cross on the computer screen indicating the movement of the platform. The assessed person tries to keep this sign on the screen in the center for 30 seconds. At the end of the test, the device calculates a balance score.
Evaluation of Gait Parameters | 4 weeks
  In the gait analysis system, the results are transferred to the computer via bluetooth with the analysis port attached to the patient's L5-S1 level. After walking, the resulting reports are automatically generated.

CONTACTS AND LOCATIONS:
Overall Officials: Gulsum Tikac, MSc Pt, Principal Investigator — Pamukkale University; Filiz Altuğ, Prof Dr, Study Director — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No